CLINICAL TRIAL: NCT01173666
Title: Renal Artery Stenosis in Coronary Artery Disease: Medical Therapy Versus Medical Therapy Plus Renal Artery Stenting in Preventing Cardiac and Renal Outcomes. The Rationale and Study Design of a Prospective,Randomized Trial: the RASCAD Study
Brief Title: Stenting of Renal Artery Stenosis in Coronary Artery Disease Study
Acronym: RASCAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Collaborators: Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government)
Responsible Party: Carmelita Marcantoni, M.D., Division of Nephrology, Cannizzaro Hospital, Catania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC-1
Record Dates: First submitted 2010-07-30; First posted 2010-08-02 (Estimated); Last update posted 2010-08-02 (Estimated); Status verified 2010-07

CONDITIONS: Renal Artery Stenosis; Left Ventricular Hypertrophy
Keywords: RAS; LVMI; Renal revascularization
MeSH Terms: conditions — Renal Artery Obstruction; Hypertrophy, Left Ventricular | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug therapy (Placebo Comparator): Patients will be treated by standard medical therapy.
  Interventions: Drug: Medical therapy
- Drug therapy + stenting angioplasty (Experimental): Patients will be treated by standard medical therapy + stenting angioplasty of renal artery.
  Interventions: Procedure: stenting angioplasty plus medical therapy

INTERVENTIONS:
Procedure: stenting angioplasty plus medical therapy — Patients will be treated by stenting angioplasty of renal artery plus medical therapy. Medical therapy is based on antihypertensive, statin or antiplatelet drugs according to clinical indications.
  Arms: Drug therapy + stenting angioplasty
Drug: Medical therapy — Patients will be treated by standard medical therapy. Medical therapy is based on antihypertensive, statin or antiplatelet drugs according with clinical indications.
  Arms: Drug therapy

SUMMARY:
The Stenting of Renal Artery Stenosis in Coronary Artery Disease (RASCAD) study is a randomized controlled trial designed to evaluate the effect of renal artery stenting+medical therapy versus medical therapy alone on left ventricular mass progression and cardiovascular morbidity and mortality in patients affected by coronary artery disease and renal artery stenosis.

DETAILED DESCRIPTION:
Patients with renal artery stenosis (RAS) have high frequency of alterations of left ventricular mass and function. Whether renal revascularization can improve cardiac function and structure in patients with RAS is not known.

The Stenting of Renal Artery Stenosis in Coronary Artery Disease (RASCAD) study was planned to test whether renal artery revascularization, compared with medical therapy, affects left ventricular hypertrophy progression and clinical outcomes in a high-risk population such as patients with evidence of coronary artery disease and RAS.

Incidental patients affected by ischemic heart disease,undergoing cardiac catheterization at a single institution, are also evaluated for the presence of RAS by renal angiography at the end of coronarography. Patients with RAS >50% and ≤80% are randomly assigned to stenting angioplasty plus medical therapy (angioplasty group) or to medical therapy alone (drug therapy group)and followed up. Patients, randomly assigned to the angioplasty group, are revascularized by stenting. All randomized patients receive antihypertensive, statin or antiplatelet drugs according to clinical indications. The planned duration of follow-up is 5 years.

The health profile of patients is described in full at study entry. Cardiovascular events (AMI, re-PTCA, cardiac heart failure, stroke,peripheral vascular disease),death, hospitalizations and medications are carefully registered throughout the study.

Standard echocardiography and renal ultrasound studies are performed at baseline and repeated every year. Echocardiography is performed following American Society of Echocardiography guidelines. LV mass is estimated using the Devereux formula and indexed to body surface area.

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease
* angiographic diagnosis of atherosclerotic RAS >50% and ≤80%

Exclusion Criteria:

* Atherosclerotic RAS>80%
* RAS secondary to fibromuscular dysplasia
* AMI
* single functioning kidney and/or sCr >4 mg/dl
* severe aortic valve stenosis
* aortic aneurism necessitating surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2006-04; Primary Completion 2011-04 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Mass (LVMI, g/m2) changes | 1 year
  Intervention in patients with RAS was hypothesized to produce a reduction in LVMI in a range between 5 to 10 g/m2. By using a 2-sided 2-sample t-test, it was calculated that a sample size of 168 patients (84 in the revascularization arm and 84 in the medical management arm) provides a 80% power to detect as significant (p<0.01) a difference of -4.0 g/m2 between patients in the revascularization arm (expected change in LVMI: -9.2 ± 7.9 g/m2) and those in the medical management arm (expected change in LVMI: -5.2 ± 5.9 g/m2).

SECONDARY OUTCOMES:
Cardiovascular mortality and morbidity | 5 years
Progression of renal function | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carmelita Marcantoni, M.D., Principal Investigator — Nephrology Division, Cannizzaro Hospital, Catania, Italy
Locations (1):
- Cardiology Division, University of Catania, Azienda Policlinico-Vittorio Emanuele, Catania, Italy

REFERENCES:
- [Background] Wright JR, Shurrab AE, Cooper A, Kalra PR, Foley RN, Kalra PA. Left ventricular morphology and function in patients with atherosclerotic renovascular disease. J Am Soc Nephrol. 2005 Sep;16(9):2746-53. doi: 10.1681/ASN.2005010043. Epub 2005 Jul 27. PMID 16049071
- [Background] Zeller T, Rastan A, Schwarzwalder U, Muller C, Frank U, Burgelin K, Sixt S, Schwarz T, Noory E, Neumann FJ. Regression of left ventricular hypertrophy following stenting of renal artery stenosis. J Endovasc Ther. 2007 Apr;14(2):189-97. doi: 10.1177/152660280701400211. PMID 17488176
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Marcantoni C, Zanoli L, Rastelli S, Tripepi G, Matalone M, Mangiafico S, Capodanno D, Scandura S, Di Landro D, Tamburino C, Zoccali C, Castellino P. Effect of renal artery stenting on left ventricular mass: a randomized clinical trial. Am J Kidney Dis. 2012 Jul;60(1):39-46. doi: 10.1053/j.ajkd.2012.01.022. Epub 2012 Apr 10. PMID 22495466